CLINICAL TRIAL: NCT02916095
Title: Evaluation Kanitinib Treatment of Recurrent or Metastatic Malignant Solid Tumors Safety, Tolerability and Pharmacokinetic Open, Dose Escalation Phase I Clinical Study
Brief Title: Kanitinib in Treating Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Beijing Konruns Pharmaceutical Co., Ltd. (Industry)
Collaborators: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KNTN-I-01
Record Dates: First submitted 2016-08-25; First posted 2016-09-27 (Estimated); Last update posted 2020-09-03 (Actual); Status verified 2020-09

CONDITIONS: Solid Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Kanitinib (Experimental): Subjects will be enrolled in cohorts at different dose levels in order to evaluate the safety,tolerability and determine the maximum tolerated dose and recommended phase II dose of kanitinib.
  Interventions: Drug: Kanitinib

INTERVENTIONS:
Drug: Kanitinib — Oral administration of Kanitinib tablets.
  Other Names: CX1003

SUMMARY:
The purpose of this study is to evaluate the safety , tolerability, pharmacokinetics of Kanitinib and determine the optimal dose in patients with recurrent or metastatic solid tumors.

DETAILED DESCRIPTION:
Evaluation of recurrent or metastatic solid tumor patients on Kanitinib single dose and continuous multiple dose safety and tolerability, and to determine the maximum tolerated Connie imatinib dose (MTD) or the phase II trial recommended dosage.

ELIGIBILITY:
Inclusion Criteria:

* 18 years to 65 years old, both genders
* patients (recruited in dose-escalation stage and dose-expansion stage) with recurrent or metastatic solid tumors are confirmed by histology staining. medullary thyroid carcinoma, radioactive iodine resistant differentiated thyroid cancers, renal cell carcinomas, lung cancers, liver cancers, gastric cancers and prostate cancers are priority selections.
* Patients are not response to standard therapy or not able to tolerate standard therapy.
* Have measurable tumor lesion (evaluated by RECIST1.1 criteria.)
* Vital organs without seriously abnormality
* With Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Expected survival time estimated to be at least 12 weeks
* Competent to comprehend, sign, and date an approved informed consent form

Exclusion Criteria:

* Absolute neutrophil count (ANC) < 1.5 x 109 / L or platelet < 100 x 109 / L or hemoglobin < 9 g/dL (refer to the normal reference range in clinical trial center).
* Total bilirubin > 1.5×the upper limit of normal range (ULN).
* Aspartate aminotransferase （AST）and/or Alanine transaminase（ALT）and/or Alkaline phosphatase(ALP) >1.5xULN without liver metastases ; AST and/or ALT and/or ALP levels ≥5xULN with liver metastases .
* Serum creatinine >1.5xULN.
* The porthrombin international normalized ratio (INR)and activated partial thromboplastin time (aPPT) >1.5xULN
* Receive chemotherapy (within 2 weeks with short half-time TKIs reagents), hormonal therapy,radiation therapy, biologics therapy or immunotherapy (within 6 weeks with nitrosoureas or mitomycin) 4 weeks prior to enrolment, except for:

  * Gonadotrophin releasing hormone (GnRH) therapy for prostate cancer
  * Hormone-replacement therapy or oral contraceptives
* Adverse events from prior anti-cancer therapy that have not resolved to Grade ≤ 1, except for alopecia.
* Brain metastasis or spinal cord compression not definitively treated with surgery and/or radiation therapy, or Brain metastases or spinal cord compression received treatments but without image evidence of showing stability ≥ 14 days.
* prior or presence of other malignancies ,with the exception of previously treated stage I B or lower grade cervical cancer， noninvasive basal cell or squamous cell cancer, breast cancer with complete remission (CR) > 10 years ,melanoma with CR > 10 years or other malignant tumors with CR > 5 years.
* Any of the following gastrointestinal disease:

  * Active gastric and duodenal ulcer or intestinal obstruction;
  * History of abdominal fistula, gastrointestinal perforation or abdominal abscess, or active digestive tract bleeding.
* Presence of hemorrhage (hemoptysis) or thrombosis disease，or currently receiving treatment with warfarin, aspirin, low molecular weight heparin (LMWH), or any other anti-platelet drugs(low dose of above mentioned drugs for prophylaxis are allowed)
* History of nephrotic syndrome.
* Patients with active infection, mental disorders or other serious nonmalignant diseases, such as congestive heart failure or unstable angina within 3 months prior to study entry, myocardial infarction or stroke within six months prior to study entry, serious arrhythmia; or those who receive therapeutical dose of anti-hypertension drugs with systolic blood pressure ≥160 mmHg or diastolic blood pressure≥100 mmHg （measured at least twice）.
* Receive surgery(including minimally invasive biopsy, open biopsy or major injuries) within 30 days, or unhealed surgical incision, ulcer , fractures, tooth extraction or other dental surgery with open wounds.
* Inability to take oral medication, prior surgical procedures or serious gastrointestinal disorders such as dysphagia and other disease that may affect drug absorption in the opinion of the investigator.
* With clinical significance of liver disease history, including viral or other hepatitis , or cirrhosis.
* Known human immunodeficiency virus infection.
* Pregnant or lactating women or those who do not take contraceptives, including men.
* Inability to comply with study and follow-up procedures
* Involved in other clinical trials < 30 days prior to enrollment.
* Any other diseases, metabolic dysfunction, abnormal physical examination findings, or clinical laboratory findings. According to investigators' judgment, patients has certain diseases or conditions are not suitable for using study drug, or affect the interpretation of the results of study, or high risk patients

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2020-01 (Actual); Study Completion 2020-07 (Actual)

PRIMARY OUTCOMES:
Adverse events accessment, changes of physical signs, laboratory examination and 12-lead electrocardiogram. | 2 year
  The safety and tolerability will be assessed according to NCI CTC AE V4.03, other safety indexes include adverse events, changes of physical signs, laboratory examination (hematology, blood biochemistry, urine routine, etc.) and a 12-lead electrocardiogram.
Maximum tolerated dose (MTD) and/or recommended Phase 2 dose (RP2D) of Kanitinib in subjects with advanced solid tumors | 2 year

CONTACTS AND LOCATIONS:
Overall Officials: Yuankai Shi, Dr, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (1):
- Cancer Institute and Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No